CLINICAL TRIAL: NCT01287013
Title: Prospective Randomized Trial Comparing Navigation With Xperguide vs. Conventional Methods During Percutaneous Image Guided Procedures
Brief Title: Comparing Xperguide vs. Conventional Methods During Percutaneous Image Guided Procedures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Investigator left NIH
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 110082; 110082 (Other: NIH Clinical Center)
Record Dates: First submitted 2011-01-25; First posted 2011-02-01 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-10

CONDITIONS: Infection; Cancer; Neoplasm; Empyema; Granuloma
Keywords: Image Guided Procedures; Xperguide CT; Electromagnetic Tracking; Navigation; Image Guided Procedure; Cancer; Granuloma
MeSH Terms: conditions — Infections; Neoplasms; Empyema; Granuloma | interventions — Cone-Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cone Beam CT (Other): Procedure performed with Xperguide cone-beam Computed Tomography (CT) navigation
  Interventions: Device: Cone-beam computed tomography (CT)
- Conventional CT (Other): Procedure performed with Conventional Computed Tomography (CT) image guidance
  Interventions: Device: Conventional Computed Tomography (CT)

INTERVENTIONS:
Device: Cone-beam computed tomography (CT) — Imaging
  Other Names: XperCT (Philips, Best); XperGuide CT
  Arms: Cone Beam CT
Device: Conventional Computed Tomography (CT) — Imaging
  Other Names: Conventional CT (Philips)
  Arms: Conventional CT

SUMMARY:
Background:

- Procedures that use medical tools in or near a possible abnormality in the body often use computed tomography (CT) scans to locate the abnormality and guide the path that a needle will take to collect a sample of tissue. Xperguide and electromagnetic (EM) tracking are two new procedures being studied to help guide the needle. Xperguide is software that uses CT images to help the doctor choose the needle path. EM tracking uses special medical tools with miniature coils that act like a Global Positioning Satellite (GPS) device to show the location of the needle in the body. Xperguide and EM tracking have been used in humans and have good results, but they have not been compared with each other and regular CT to determine whether they are better than the standard approach.

Objectives:

- To compare the results of Xperguide, electromagnetic tracking, and regular computed tomography during a guided percutaneous procedure.

Eligibility:

- Individuals at least 18 years of age who are required to have a CT-guided percutaneous procedure.

Design:

* Participants will be screened with a physical examination and medical history, and the results of any previous imaging studies will be examined before study enrollment.
* After a pilot phase, the study will involve two phases to compare the results of the different procedures. The first phase will involve comparing Xperguide to CT, and the second will involve comparing Xperguide to EM tracking.
* Phase 1 participants will be assigned to one of two procedure groups: Group 1 will have Xperguide, and Group 2 will have regular CT. Participants who are scheduled to have repeated procedures (like a biopsy before and after chemotherapy) will be randomized for the first procedure and the second procedure will be done using the other method.
* Phase 2 participants will be assigned to one of two procedure groups: Group 1 will have Xperguide, and Group 2 will have EM tracking. Participants who are scheduled to have repeated procedures (like a biopsy before and after chemotherapy) will be randomized for the first procedure and the second procedure will be done using the other method.
* Standard post-procedure followup care will be given after the study procedure is completed.

DETAILED DESCRIPTION:
PR(SqrRoot) CIS

This is a phase II prospective randomized trial comparing a novel navigation method, Xperguide to conventional CT and electromagnetic tracking (EM) during percutaneous image guided procedures. Xperguide is a navigation tool that utilizes a cone beam CT (CBCT) obtained in the angiography suite overlaid on fluoroscopy for needle guidance during image guided procedures. The needle entry point and path are planned on the CBCT and the determined path is overlaid on fluoroscopy image for real time guidance.

SPECIFIC AIMS/OBJECTIVES

1. The primary aims are:

   a. Pilot trial:

   i. To familiarize operators with outcome measures allowing for fair comparison in the subsequent study

   b. Main trial will have 2 phases with similar outcomes criteria and aims (below):

   i. comparing Xperguide to conventional imaging (superiority design):

ii. comparing Xperguide to EM tracking (equivalence design):

1. To compare the accuracy of final device tip position and path (vector)
2. To compare the number of repositioning maneuvers
3. To compare the radiation dose
4. To compare rates of definitive pathological diagnosis and response rate per EASL criteria for ablations

METHODS/METHODOLOGY

For non-vascular image guided interventions, patients undergoing biopsies and ablations procedures requiring CT guidance are eligible for inclusion and randomization. An initial pilot study will be done in which each operator will perform at least 5 cases using Xperguide completing the case report forms. This will ensure experience with outcome measures and fair comparison in the subsequent study. Once one of the operators reaches the minimal required cases, the main trial will begin for that operator. However every other operator must each complete the minimal number of cases with the case report forms to enroll patients in the main trial. Initially, we will compare Xperguide with conventional CT with several cohorts of patients mainly: lung biopsies, and ablations, kidney biopsies/ablations and other abdominal biopsies/ ablations. In ablations of large lesions, Xperguide composite ablation software can provide input on the expected ablation zones. Each probe will be positioned in the same manner as any biopsy needle following steps described in section 4. If this specific composite ablation module of the

software is not commercially released and FDA cleared at the time of the study, then this software will only be used on protocol to help the physician determine ideal needle positioning for complete ablation. Once consent is obtained the participant is randomized to either conventional imaging or Xperguide. In addition, if it is known that the patient is participating in a trial which requires a repeat (paired, pre and post treatment) procedure of the same site, then the randomization will determine which modality is used for guidance at the first visit and the other modality will automatically be used for the second procedure. In these cases, if the patient gives consent they will be randomized to one of two categories:

1. Xperguide for the initial procedure and conventional CT for the 2nd procedure
2. Conventional CT for the initial procedure and Xperguide for the 2nd procedure

Then in the second phase of the trial, Xperguide will be compared to EM tracking for biopsies and ablations requiring CT guidance, in an equivalence study. Once consent is obtained, the participant will be randomized into EM tracking or Xperguide. The patients would be divided into different cohorts depending on the anatomic site of the interventions i.e. lung, kidney, liver and other abdomen. If the patients are participating in a trial requiring paired procedures (i.e. pre and post treatment), the randomization will determine which modality is used for the initial procedure and the other modality will be used for the second procedure. In summary there will be two potential categories:

1. EM tracking for the initial procedure and Xperguide for the 2nd procedure
2. Xperguide for the initial procedure and EM tracking for the 2nd procedure

If a patient has a lesion that is only visible on PET-CT/MR, or demonstrates heterogenous PET-CT/MR uptake, there will be a separate cohort of PET-CT/MR guided biopsies and ablations using Xperguide vs EM tracking. There is also the need for a cohort for ablations with complimentary use of ultrasound at the discretion of the operator in order to conform to our standard of care at the NIH.

ELIGIBILITY

Subjects are eligible if:

1. they are over 18 years of age
2. they are scheduled for image guided procedure
3. the lesion is not superficial (deeper than 3cm)

Subjects are excluded if:

1. they have an altered mental status that precludes understanding or consenting for the procedure
2. they are unable to hold reasonably still on a procedure table for the length of the procedure
3. they are unable to hold their breath if the procedure will be performed with conscious sedation and without general anesthesia
4. their gross body weight is over 375 pounds which the upper limit of the CT and

angiography tables

REQUIRED SAMPLE SIZE

A pilot study will be performed to ensure operator experience with Xperguide and EM tracking, for fair comparison. In the pilot study each operator must perform 5 cases with Xperguide completing the case report forms. There are 5 potential operators therefore a maximum of 25 patients (if all 5 operators participate to the fullest).

The first phase of the main trial comparing Xperguide with conventional CT was powered (for sample size) with a standard superiority design aimed to statistically establish that Xperguide is better than conventional CT (defined as requiring fewer needle repositioning efforts). These calculations yield a total sample size of 60 patients with 20 patients per anatomical site.

For the second phase of the trial comparing Xperguide to EM tracking, a two sided equivalence design (based on accuracy and number of needle repositioning) was used for sample size considerations, and yielded 192 patients. Therefore 16 patients per modality per anatomical site will be randomized with two additional cohorts for PET-CT/MR procedures and composite ablations.

Number of Participants: 277

Recruitment Time Frame: 4 years

Number of sites: 1

Type of Study: prospective randomized clinical trial after an initial pilot period

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. they are over 18 years of age
  2. they are scheduled for image guided procedure
  3. the lesion is not superficial (deeper than 3 cm)

EXCLUSION CRITERIA:

1. patients with an altered mental status that precludes understanding or consenting for the procedure
2. patients unable to hold reasonably still on a procedure table for the length of the procedure
3. patient unable to hold their breath if the procedure will be performed with conscious sedation and without general anesthesia
4. patient with a gross body weight over 375 pounds (upper limit of the CT and angiography tables)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradford Wood, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carrafiello G, Mangini M, De Bernardi I, Fontana F, Dionigi G, Cuffari S, Imperatori A, Lagana D, Fugazzola C. Microwave ablation therapy for treating primary and secondary lung tumours: technical note. Radiol Med. 2010 Sep;115(6):962-74. doi: 10.1007/s11547-010-0547-7. Epub 2010 Mar 29. English, Italian. PMID 20352357
- [Background] Racadio JM, Babic D, Homan R, Rampton JW, Patel MN, Racadio JM, Johnson ND. Live 3D guidance in the interventional radiology suite. AJR Am J Roentgenol. 2007 Dec;189(6):W357-64. doi: 10.2214/AJR.07.2469. PMID 18029850
- [Background] Spelle L, Ruijters D, Babic D, Homan R, Mielekamp P, Guillermic J, Moret J. First clinical experience in applying XperGuide in embolization of jugular paragangliomas by direct intratumoral puncture. Int J Comput Assist Radiol Surg. 2009 Nov;4(6):527-33. doi: 10.1007/s11548-009-0370-6. Epub 2009 Jun 13. PMID 20033329
- [Result] Abi-Jaoudeh N, Fisher T, Jacobus J, Skopec M, Radaelli A, Van Der Bom IM, Wesley R, Wood BJ. Prospective Randomized Trial for Image-Guided Biopsy Using Cone-Beam CT Navigation Compared with Conventional CT. J Vasc Interv Radiol. 2016 Sep;27(9):1342-1349. doi: 10.1016/j.jvir.2016.05.034. Epub 2016 Jul 25. PMID 27461586
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-CC-0082.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period = 2/4/2011 - 5/15/2014 Recruitment location = Interventional Radiology Clinic, Department of Radiology and Imaging Sciences, Clinical Center, NIH
Pre-assignment Details: The PILOT Arm of the study was done prior to enrolling participants in the main phase of the study. PILOT Participants were enrolled to familiarize operators with performing Xperguide procedures. Participants enrolled in the PILOT Arm were not randomized to either the Cone Beam CT or Conventional CT Arms and not included in the analysis.
Groups:
- PILOT: Procedures performed with Xperguide without randomization to familiarize operators.
Period: Overall Study
Arm/Group | Cone Beam CT | Conventional CT | PILOT
Started | 32 | 34 | 21
Completed | 29 | 29 | 0
Not Completed | 3 | 5 | 21
Not completed — Non-evaluable | 3 | 5 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cone Beam CT | Conventional CT | PILOT | Total
Number analyzed (Participants) | 32 | 34 | 21 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 1
  Between 18 and 65 years | 25 | 25 | 8 | 58
  >=65 years | 7 | 9 | 12 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 8 | 4 | 30
  Male | 14 | 26 | 17 | 57

OUTCOME MEASURES:

1. Primary Outcome: Comparing the Accuracy of Final Device Tip Position
Description: To compare the accuracy of the biopsy needle between the software guidance and conventional CT. The accuracy of the needle position was calculated in millimeters by using the difference between the x,y,z coordinates of the tip of the actual needle before specimen collection. Actual and planned needle paths were compared using coordinates and measured in millimeters.
Time Frame: 1 hour
Population: Participants enrolled in the PILOT Arm were not randomized to the Cone Beam CT or Conventional CT Arms and were not included in the analysis. PILOT Participants were enrolled to familiarize operators with performing Xperguide procedures.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Cone Beam CT | Conventional CT
Number analyzed (Participants) | 29 | 29
mm | 4.9 (4.1) | 12.2 (8.1)
Statistical Analysis 1: Comparison: Cone Beam CT vs Conventional CT; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Accuracy of Final Device Path (Vector)
Description: Comparing the accuracy of the path the biopsy needle took to get to the site
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Convetional CT: Procedure performed with Conventional Computed Tomography (CT) image guidance
Arm/Group | Cone Beam CT | Convetional CT
Number analyzed (Participants) | 29 | 29
mm | 8.8 (5.4) | 28.3 (20.5)
Statistical Analysis 1: Comparison: Cone Beam CT vs Convetional CT; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Radiation Doses Between Xperguide and Conventional CT
Description: Comparing radiation doses to determine if there is a change in the dose between the two interventions
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Cone Beam CT | Conventional CT
Number analyzed (Participants) | 29 | 29
mGy | 53.3 (33.3) | 75.4 (62.6)
Statistical Analysis 1: Comparison: Cone Beam CT vs Conventional CT; Test type: Other; p < 0.04, t-test, 2 sided

4. Secondary Outcome: Compare the Number of Repositioning Maneuvers
Description: To compare the number of times the needle must be repositioned during the guidance of the needle to the biopsy.
Time Frame: 1 hour
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of repositioning maneuvers
Arm/Group | Cone Beam CT | Conventional CT
Number analyzed (Participants) | 29 | 29
number of repositioning maneuvers | 0.3 (0.5) | 1.9 (2.3)
Statistical Analysis 1: Comparison: Cone Beam CT vs Conventional CT; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

5. Secondary Outcome: Rates of Definitive Pathologic Diagnosis
Description: Definitive pathologic diagnosis was defined as an adequate specimen as judged by the pathologist and a diagnosis confirmed by surgery or clinical follow-up.
Time Frame: 1 hour
Population: as for outcome 1
Measure: Number; unit: percent of accuracy
Arm/Group | Cone Beam CT | Conventional CT
Number analyzed (Participants) | 29 | 29
percent of accuracy | 93.9 | 90.9
Statistical Analysis 1: Comparison: Cone Beam CT vs Conventional CT; Test type: Superiority or Other; p = 0.67, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 1 day
Groups:
- Pilot Arm: Pilot participants were enrolled to familiarize operators with performing Xperguide procedures.
Arm/Group | Cone Beam CT | Conventional CT | Pilot Arm
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/29 | 1/29 | 0/21
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cone Beam CT (N=29) | Conventional CT (N=29) | Pilot Arm (N=21)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Grade 3. Possibly related to research (procedure). Patient was hospitalized for 3 days for a small left apical pneumothorax increased since immediate post lung biopsy verified by chest CT. A chest tube had to be placed in IR after the biopsy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes